CLINICAL TRIAL: NCT02840071
Title: Acceptance and Commitment Therapy for Individuals With Head and Neck Cancer Experiencing Psychological Distress: A Hermeneutic Single-Case Efficacy Design
Brief Title: ACT for Distress in Head and Neck Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16067
Record Dates: First submitted 2016-07-12; First posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Psychological therapy.
  Interventions: Other: Psychological therapy

INTERVENTIONS:
Other: Psychological therapy — Acceptance and commitment therapy is a third-wave cognitive behavioural therapy. The aim of ACT intervention is to increase a person's psychological flexibility by enabling them to change their relationship with distressing cognitions (acceptance) and doing things that are personally meaningful to them (commitment). The ACT model does not focus on distress reduction, although this is a secondary consequence of acceptance and commitment. This is targeted through the six core processes: present moment awareness, cognitive defusion, acceptance, self-as-context, values and committed action which means taking effective action, guided by the identified values. The intervention will involve six 1.5 hourly individual sessions.

SUMMARY:
Title: Acceptance and Commitment therapy for Individuals with Head and Neck Cancer Experiencing Psychological Distress.

Head and neck cancer (HNC) patients are particularly vulnerable to experiencing psychological distress . The current guidelines from the National Institute of Health and Care Excellence are that cognitive-behavioural therapy (CBT) is to be offered to adults with a long-term physical health condition experiencing anxiety and depression. CBT has been shown to have several inadequacies for individuals with physical health conditions such as cancer. Acceptance and commitment therapy (ACT) takes an alternative approach to CBT, aiming to change a person's interaction with their thoughts rather than suppress or alter thought content. Although studies indicate encouraging findings for the effectiveness of ACT for individuals with breast cancer; the HNC- transfer-ability of findings is yet untested, and there is a need to evaluate the replicability of ACT effects in people living with HNC, given the unique challenges inherent to the disease and its treatment.

This study aims to inform clinical practise by using a hermeneutic single-case efficacy design (HSCED) to answer the following questions:

1. Is there evidence of psychological change after the introduction of the ACT intervention?
2. If present, are the changes attributable to (a) ACT components, (b) common factors, and/or (c) non-therapeutic factors?

The study will involve recruiting three adults with HNC from specialist HNC psychology services. Each participant will have six individual sessions of ACT and complete various process and outcome questionnaires during sessions. Following the intervention, participants will have a semi-structured interview where their views of the therapy and any changes made will be explored. Two outcome measures will be posted to participants at 1-month and 3-month post intervention.

DETAILED DESCRIPTION:
This study aims contribute to the theoretical literature on acceptance and commitment therapy (ACT) as well as the processes of psychological change for patients with head and neck cancer (HNC). Unlike some other cancer sites, the physical and emotional impact of living with HNC can be detrimental to the fundamental aspects of an individual's life (such as breathing, eating, hearing), and also cause significant changes to physical appearance. This forms the basis for specialised research of HNC patients. There is a tendency within the current cancer literature towards researching and understanding and other types of cancer or grouping HNC patients into heterogeneous cancer samples, leaving an evident gap of knowledge. Studies that have assessed the effectiveness of ACT mirror this trend, using either breast cancer or heterogeneous cancer samples.

Employing a single-case method with both quantitative and qualitative components will give a more precise understanding of the processes within ACT that are helpful and most importantly, why. This may have direct implications for informing the on-going practice of professionals working therapeutically using ACT, enabling them to refine interventions and focal principles. In support of this, a recent review of ACT interventions concluded that although efficacy of ACT is probable, there is a lack of knowledge of how it works. Single-case research is a pragmatic first step in exploring the efficacy of ACT for HNC patients and increasing understanding of the potential mechanisms of change. A Hermeneutic Single Case Efficacy Design for three participants will be used. This is a legalistic single case study method which allows the assessment of intervention effects in single therapy cases within a naturalistic clinical context. It uses a mixture of qualitative(change interview) and quantitative methods (questionnaires) to create a set of evidence that allows detection of causal links between therapy process and outcome.

In order to minimise the risk of coercion, a member of the patients care team (Clinical Psychologist) will be the first point of contact for potential participants, introducing waiting-list patients to the research and giving them the information sheet if they verbally indicate interest. After reading the information sheet, if they verbally agree to continue with the research, they will be put into contact with the researcher who will answer any additional questions, ensuring that the person has sufficient time to consider participating or not. Written informed consent will be collected from each participant before they undergo any intervention related to the study. One copy of this will be kept by the participant, one will be kept by the researcher, and a third will be retained in the patient's hospital records.

Informed consent will be gained in accordance with the Research Ethics Committee (REC) guidance, and Good Clinical Practice (GCP) and any other regulatory requirements that might be introduced. The researcher and the participant will both sign and date the informed consent form before the person can participate in the study. The researcher will emphasise to them that consent regarding study participation is entirely voluntary and may be withdrawn at any time without penalty or affecting their care. For example, if the patient withdraws from the study, they will return to the point of the psychological therapy waiting list that they were taken from, therefore not affecting the length of time they have to wait to see a therapist. There will be no monetary incentive to take part in the research, reducing the risk of coercion.

This research aims to use a sample most representative of individuals in clinical practice, therefore site and stage of HNC does not feature the inclusion criteria. The GAD-7 (generalised anxiety disorder) and PHQ-9 (patient health: depression) questionnaires will be used using 'caseness' thresholds for anxiety and/or depression as these are widely used and the current screening method for most psychology therapy services.

In order to ensure confidentiality, identification code numbers will be assigned to correspond to treatment data. All study researchers will endeavour to protect the rights of the participants to privacy and will adhere to the Data Protection Act, 1998. Only the minimum required information for the purposes of the study will be collected. Participant information will be held securely, in a locked room, or locked cupboard or cabinet. Access to the information will be limited to the study staff and investigators. Computer held data including the study database will be held securely and password protected. All data will be stored on a secure dedicated web server. Access will be restricted by user identifiers and passwords (encrypted using a one way encryption method). Information about the study in the participant's medical records / hospital notes will be treated confidentially in the same way as all other confidential medical information.

There are no likely risks for participants taking part in the study, other than iatrogenic effects that are a possibility with any psychological therapy. These include: increased insight into difficulties causing an increase in psychological distress and psychological discomfort talking about physical and psychological distress. These risks would be monitored throughout therapy using the standardised measures and clinical observations. If these risks appear to be occurring, the chief investigator will be notified and the service safeguarding protocols will be followed, as patients will remain under the HNC psychology service during the course of the research.

There are several potential benefits to participants taking part in this research as suggested by the ACT cancer literature: reduced psychological distress, increased psychological flexibility and improved quality of life. As the researcher is also the therapist, any potential conflict of interest will be managed by using fortnightly clinical supervision with a psychologist, having a random 20% of the the audio recorded sessions viewed by a specialist ACT psychologist and having an independent researcher to carry out the change interview.

After receiving informed consent the study procedure will be as follows:

* Trainee Clinical Psychologist (researcher) will deliver an ACT intervention using the Better Living with Illness Protocol. This will involve six 1.5 hour sessions at a clinic room at the relevant hospital site (King's Mill/City). Sessions will be audio recorded.
* Two process measures (questionnaires) will be given at the end of each session. Two outcome measures will be given at the end of first and last session.
* Upon completion of the intervention, each participant will individually meet with an independent researcher (Trainee Psychologist on the Doctorate of Clinical Psychology, University of Nottingham) at King's Mill Hospital for a 30 minute semi-structured interview. This will follow the Client Change Interview Protocol and Helpful Aspects of Therapy framework. The aim of this is to collect qualitative information about the clients view of any changes noticed over the duration of the therapy and the attributions for these changes.
* Finally, participants will be posted two outcome measures at 1-month post intervention and 3-month post intervention.

ELIGIBILITY:
Inclusion Criteria:

Participants taking part must:

* Be above the age of 18
* Have capacity to give informed consent (assessed by the clinical psychologist within the service)
* Able to understand and speak the English language
* Have a diagnosis head and neck cancer
* Experiencing psychological distress (assessed using anxiety and depression screening tools)
* Have the ability to attend relevant hospital for study participation

Exclusion Criteria:

* N/A see above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change in psychological flexibility assessed using the Acceptance and Action Questionnaire (AAQ-II) | up to 18 weeks
  The primary goal of ACT is increasing psychological flexibility by enabling a person to change their relationship with distressing cognitions (acceptance) and do things that are personally meaningful to them (commit). The primary outcome will be an assessment of whether change has occurred using process measures (acceptance and action questionnaire: AAQ-II).
Change in psychological flexibility assessed using the Problem Questionnaire (PQ) | up to 18 weeks
  Changes in the problem questionnaire (PQ) (administered pre and post intervention) will also be used as an indirect measure of change in psychological flexibility. This measure consists of up to 10 unique problem statements that the individual has, rated on a 7-point likert scale. Significant reductions in these ratings would indicate an increase in psychological flexibility.

SECONDARY OUTCOMES:
Depression assessed by PHQ-9 questionnaire | up to 18 weeks
  In line with the theoretical underpinnings of ACT, a secondary consequence of an increase in psychological flexibility is a reduction in psychological distress. The study will measure changes in psychological distress (depression) using PHQ-9 (patient health: depression questionnaire). A clinical caseness score (10 or above) is a threshold for clinical levels of depression. Analysis to identify statistically reliable change (pre and post intervention and follow up) will be carried out.
Anxiety assessed by GAD-7 questionnaire | up to 18 weeks
  In line with the theoretical underpinnings of ACT, a secondary consequence of an increase in psychological flexibility is a reduction in psychological distress. The study will measure changes in psychological distress (anxiety) using GAD-7 (generalised anxiety disorder questionnaire). A clinical caseness score (8 or above) is a threshold for clinical levels of anxiety. Analysis to identify statistically reliable change (pre, post intervention and follow-up) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schroder, Psychology, Principal Investigator — University of Nottingham
Locations (2):
- United Kingdom (2):
  - City Hospital, Nottingham, Notitnghamshire
  - King's Mill Hospital, Mansfield, Nottinghamshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elliott R. Hermeneutic single-case efficacy design. Psychother Res. 2002 Mar 1;12(1):1-21. doi: 10.1080/713869614. PMID 22471329
- [Background] Frampton M. Psychological distress in patients with head and neck cancer: review. Br J Oral Maxillofac Surg. 2001 Feb;39(1):67-70. doi: 10.1054/bjom.2000.0547. PMID 11178847
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724
- [Background] Hulbert-Williams NJ, Storey L, Wilson KG. Psychological interventions for patients with cancer: psychological flexibility and the potential utility of Acceptance and Commitment Therapy. Eur J Cancer Care (Engl). 2015;24(1):15-27. doi: 10.1111/ecc.12223. Epub 2014 Aug 6. PMID 25100576
- [Background] Lang H, France E, Williams B, Humphris G, Wells M. The psychological experience of living with head and neck cancer: a systematic review and meta-synthesis. Psychooncology. 2013 Dec;22(12):2648-63. doi: 10.1002/pon.3343. Epub 2013 Jul 10. PMID 23840037
- [Background] Ost LG. Efficacy of the third wave of behavioral therapies: a systematic review and meta-analysis. Behav Res Ther. 2008 Mar;46(3):296-321. doi: 10.1016/j.brat.2007.12.005. Epub 2007 Dec 23. PMID 18258216
- [Background] Ost LG. The efficacy of Acceptance and Commitment Therapy: an updated systematic review and meta-analysis. Behav Res Ther. 2014 Oct;61:105-21. doi: 10.1016/j.brat.2014.07.018. Epub 2014 Aug 19. PMID 25193001
- [Background] Vilardaga R, Bricker J, McDonell M. The promise of mobile technologies and single case designs for the study of individuals in their natural environment. J Contextual Behav Sci. 2014 Apr 1;3(2):148-153. doi: 10.1016/j.jcbs.2014.03.003. PMID 24949285
- [Background] Ruiz FJ. A Review of Acceptance and Commitment Therapy (ACT) Empirical Evidence : Correlational , Experimental Psychopathology , Component and Outcome Studies. International Journal of Psychology and Psychological Therapy 10(1): 125-162, 2010